CLINICAL TRIAL: NCT00313209
Title: Effect of Roflumilast in COPD Patients Treated With Salmeterol. A 24-week, Double-blind Study With 500 μg Roflumilast Once Daily Versus Placebo. The EOS Study
Brief Title: Effect of Roflumilast on Lung Function in Chronic Obstructive Pulmonary Disease (COPD) Patients Treated With Salmeterol: The EOS Study (BY217/M2-127)
Acronym: EOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY217/M2-127; 2005-005080-28 (EudraCT Number)
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Results first posted 2011-05-19 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Roflumilast; Salmeterol; COPD; Chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Roflumilast (Active Comparator): Roflumilast 500 µg
  underlying medication: salmeterol 50 μg, twice daily, inhaled
  Interventions: Drug: Roflumilast
- Placebo (Placebo Comparator): Placebo
  underlying medication: salmeterol 50 μg, twice daily, inhaled
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast — 500 µg, once daily, oral administration in the morning
  Arms: Roflumilast
Drug: Placebo — once daily
  Arms: Placebo

SUMMARY:
The aim of the study is to compare the efficacy of roflumilast on pulmonary function and symptomatic parameters in patients with chronic obstructive pulmonary disease (COPD) during concomitant administration of salmeterol. The study duration will last up to 28 weeks. The study will provide further data on safety and tolerability of roflumilast.

ELIGIBILITY:
Main Inclusion Criteria:

* History of COPD for at least 12 months prior to baseline visit
* FEV1/FVC ratio (post-bronchodilator) ≤ 70%
* FEV1 (post-bronchodilator) between ≥ 40% and ≤ 70% of predicted

Main Exclusion Criteria:

* COPD exacerbation indicated by a treatment with systemic glucocorticosteroids and/or antibiotics not stopped at least 4 weeks prior to baseline visit

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 933 (Actual)
Dates: Start 2006-04; Primary Completion 2007-07 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (123):
- Austria (9):
  - Altana Pharma/Nycomed Investigational Site, Linz
  - Altana Pharma/Nycomed Investigational Site, Neusiedl/See
  - Altana Pharma/Nycomed Investigational Site, Perg
  - Altana Pharma/Nycomed Investigational Site, Salzburg
  - Altana Pharma/Nycomed Investigational Site, Sankt Pölten
  - Altana Pharma/Nycomed Investigational Site, Steyr
  - Altana Pharma/Nycomed Investigational Site, Vienna
  - Altana Pharma/Nycomed Investigational Site, Wiener Neustadt
  - Altana Pharma/Nycomed Investigational Site, Zwettl Stadt
- Belgium (13):
  - Altana Pharma/Nycomed Investigational Site, Arlon
  - Altana Pharma/Nycomed Investigational Site, Brussels
  - Altana Pharma/Nycomed Investigational Site, Duffel
  - Altana Pharma/Nycomed Investigational Site, Genk
  - Altana Pharma/Nycomed Investigational Site, Gilly
  - Altana Pharma/Nycomed Investigational Site, Halen
  - Altana Pharma/Nycomed Investigational Site, Jette
  - Altana Pharma/Nycomed Investigational Site, Leuven
  - Altana Pharma/Nycomed Investigational Site, Liège
  - Altana Pharma/Nycomed Investigational Site, Malmedy
  - Altana Pharma/Nycomed Investigational Site, Montigny-le-Tilleul
  - Altana Pharma/Nycomed Investigational Site, Namur
  - Altana Pharma/Nycomed Investigational Site, Veurne
- Canada (24):
  - Altana Pharma/Nycomed Investigational Site, Ajax, Ontario
  - Altana Pharma/Nycomed Investigational Site, Halifax, N.S.
  - Altana Pharma/Nycomed Investigational Site, Hamilton
  - Altana Pharma/Nycomed Investigational Site, Hamilton, Ontario
  - Altana Pharma/Nycomed Investigational Site, Laval
  - Altana Pharma/Nycomed Investigational Site, London
  - Altana Pharma/Nycomed Investigational Site, Mirabel
  - Altana Pharma/Nycomed Investigational Site, Montreal
  - Altana Pharma/Nycomed Investigational Site, Montreal, PQ
  - Altana Pharma/Nycomed Investigational Site, New Market, on
  - Altana Pharma/Nycomed Investigational Site, North Bay
  - Altana Pharma/Nycomed Investigational Site, Ontario
  - Altana Pharma/Nycomed Investigational Site, Ottawa
  - Altana Pharma/Nycomed Investigational Site, Québec
  - Altana Pharma/Nycomed Investigational Site, Regina, Saskatchewan
  - Altana Pharma/Nycomed Investigational Site, Saint John
  - Altana Pharma/Nycomed Investigational Site, Sainte-Foy, Quebec
  - Altana Pharma/Nycomed Investigational Site, Saskatoon SK
  - Altana Pharma/Nycomed Investigational Site, Sherbrooke, PQ
  - Altana Pharma/Nycomed Investigational Site, Toronto, on
  - Altana Pharma/Nycomed Investigational Site, Vancouver, BC
  - Altana Pharma/Nycomed Investigational Site, Windsor
  - Altana Pharma/Nycomed Investigational Site, Winnipeg MB
  - Altana Pharma/Nycomed Investigational Site, Woodstock
- France (15):
  - Altana Pharma/Nycomed Investigational Site, Beausoleil
  - Altana Pharma/Nycomed Investigational Site, Beuvry
  - Altana Pharma/Nycomed Investigational Site, Chauny
  - Altana Pharma/Nycomed Investigational Site, Grasse
  - Altana Pharma/Nycomed Investigational Site, Grenoble
  - Altana Pharma/Nycomed Investigational Site, Lille
  - Altana Pharma/Nycomed Investigational Site, Lyon
  - Altana Pharma/Nycomed Investigational Site, Martigues
  - Altana Pharma/Nycomed Investigational Site, Montpellier
  - Altana Pharma/Nycomed Investigational Site, Nantes
  - Altana Pharma/Nycomed Investigational Site, Nice
  - Altana Pharma/Nycomed Investigational Site, Nîmes
  - Altana Pharma/Nycomed Investigational Site, Saint-Laurent-du-Var
  - Altana Pharma/Nycomed Investigational Site, Saint-Quentin
  - Altana Pharma/Nycomed Investigational Site, Trélazé
- Germany (16):
  - Altana Pharma/Nycomed Investigational Site, Aschaffenburg
  - Altana Pharma/Nycomed Investigational Site, Bochum
  - Altana Pharma/Nycomed Investigational Site, Bonn
  - Altana Pharma/Nycomed Investigational Site, Cologne
  - Altana Pharma/Nycomed Investigational Site, Geesthacht
  - Altana Pharma/Nycomed Investigational Site, Gelnhausen
  - Altana Pharma/Nycomed Investigational Site, Großhansdorf
  - Altana Pharma/Nycomed Investigational Site, Hanover
  - Altana Pharma/Nycomed Investigational Site, Koblenz
  - Altana Pharma/Nycomed Investigational Site, Marburg
  - Altana Pharma/Nycomed Investigational Site, Saarbrücken
  - Altana Pharma/Nycomed Investigational Site, Schwetzingen
  - Altana Pharma/Nycomed Investigational Site, Sinsheim
  - Altana Pharma/Nycomed Investigational Site, Surwold
  - Altana Pharma/Nycomed Investigational Site, Witten
  - Altana Pharma/Nycomed Investigational Site, Würzburg
- Italy (14):
  - Altana Pharma/Nycomed Investigational Site, Bari
  - Altana Pharma/Nycomed Investigational Site, Bologna
  - Altana Pharma/Nycomed Investigational Site, Catania
  - Altana Pharma/Nycomed Investigational Site, Cisanello (PI)
  - Altana Pharma/Nycomed Investigational Site, Genova
  - Altana Pharma/Nycomed Investigational Site, Livorno
  - Altana Pharma/Nycomed Investigational Site, Milan
  - Altana Pharma/Nycomed Investigational Site, Pordenone
  - Altana Pharma/Nycomed Investigational Site, Roma
  - Altana Pharma/Nycomed Investigational Site, Saluzzo (CN)
  - Altana Pharma/Nycomed Investigational Site, Torino
  - Altana Pharma/Nycomed Investigational Site, Tradate (VA)
  - Altana Pharma/Nycomed Investigational Site, Verona
  - Altana Pharma/Nycomed Investigational Site, Vittorio Veneto (TV)
- Netherlands (6):
  - Altana Pharma/Nycomed Investigational Site, Alkmaar
  - Altana Pharma/Nycomed Investigational Site, Almelo
  - Altana Pharma/Nycomed Investigational Site, Eindhoven
  - Altana Pharma/Nycomed Investigational Site, Helmond
  - Altana Pharma/Nycomed Investigational Site, Schiedam
  - Altana Pharma/Nycomed Investigational Site, Zwolle
- Altana Pharma/Nycomed Investigational Sites, Cape Town, South Africa
- Spain (11):
  - Altana Pharma/Nycomed Investigational Site, Alicante
  - Altana Pharma/Nycomed Investigational Site, Barcelona
  - Altana Pharma/Nycomed Investigational Site, Elche (Alicante)
  - Altana Pharma/Nycomed Investigational Site, Fuentesnuevas, Ponferrada (León)
  - Altana Pharma/Nycomed Investigational Site, Guadalajara
  - Altana Pharma/Nycomed Investigational Site, Laredo (Cantabria)
  - Altana Pharma/Nycomed Investigational Site, Mataró, Barcelona
  - Altana Pharma/Nycomed Investigational Site, Petrer (Alicante)
  - Altana Pharma/Nycomed Investigational Site, Sabadell
  - Altana Pharma/Nycomed Investigational Site, Tarrasa (Barcelona)
  - Altana Pharma/Nycomed Investigational Site, Torrelavega (Cantabria)
- United Kingdom (14):
  - Altana Pharma/Nycomed Investigational Site, Belfast
  - Altana Pharma/Nycomed Investigational Site, Bexhill-on-Sea, East Sussex
  - Altana Pharma/Nycomed Investigational Site, Bradford
  - Altana Pharma/Nycomed Investigational Site, Bradford on Avon, Wiltshire
  - Altana Pharma/Nycomed Investigational Site, Chesterfield Derbyshire
  - Altana Pharma/Nycomed Investigational Site, Coleraine
  - Altana Pharma/Nycomed Investigational Site, Cookstown
  - Altana Pharma/Nycomed Investigational Site, East Sussex
  - Altana Pharma/Nycomed Investigational Site, Edinburgh
  - Altana Pharma/Nycomed Investigational Site, Glasgow
  - Altana Pharma/Nycomed Investigational Site, Hastings
  - Altana Pharma/Nycomed Investigational Site, Middlessex
  - Altana Pharma/Nycomed Investigational Site, Sunbury on Thames, Middlessex
  - Altana Pharma/Nycomed Investigational Site, Watford

REFERENCES:
- [Result] Fabbri LM, Calverley PM, Izquierdo-Alonso JL, Bundschuh DS, Brose M, Martinez FJ, Rabe KF; M2-127 and M2-128 study groups. Roflumilast in moderate-to-severe chronic obstructive pulmonary disease treated with longacting bronchodilators: two randomised clinical trials. Lancet. 2009 Aug 29;374(9691):695-703. doi: 10.1016/S0140-6736(09)61252-6. PMID 19716961
- [Derived] Cazzola M, Picciolo S, Matera MG. Roflumilast in chronic obstructive pulmonary disease: evidence from large trials. Expert Opin Pharmacother. 2010 Feb;11(3):441-9. doi: 10.1517/14656560903555201. PMID 20102307

RESULTS

PARTICIPANT FLOW:
Groups:
- Roflumilast: Roflumilast 500 µg, once daily, oral and salmeterol 50 µg, twice daily, inhaled
- Placebo: Placebo, once daily, oral and salmeterol 50 µg, twice daily, inhaled
Period: Overall Study
Arm/Group | Roflumilast | Placebo
Started | 466 (Includes all randomized patients who took at least one dose of the investigational drug.) | 467 (Includes all randomized patients who took at least one dose of the investigational drug.)
Completed | 359 | 385
Not Completed | 107 | 82

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Roflumilast | Placebo | Total
Number analyzed (Participants) | 466 | 467 | 933
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (8.7) | 64.9 (9.3) | 64.9 (9.0)
Gender [Count of Participants; unit: Participants]
  Female | 147 | 168 | 315
  Male | 319 | 299 | 618

OUTCOME MEASURES:

1. Primary Outcome: Pre-bronchodilator Forced Expiratory Volume in First Second (FEV1)
Description: Mean change from baseline during the treatment period in pre-bronchodilator FEV1 [L]
Time Frame: Change from baseline over 24 weeks of treatment
Population: ITT (Intention to Treat) analysis. Number of participants analyzed = number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 456 | 463
mL | 39 (9) | -10 (9)
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment of the significance level (0.05) was done as a hierarchical approach for hypotheses testing was used; Repeated measurements analysis (change from baseline over 24 weeks of treatment taking all post-randomization measurements into account); Mean Difference (Net) = 49, 95% CI 2-sided [27 to 71], Standard Error of Mean 11

2. Secondary Outcome: Post-bronchodilator FEV1
Description: Mean change from baseline during the treatment period in post-bronchodilator FEV1 [L]
Time Frame: Change from baseline over 24 weeks of treatment
Population: ITT analysis. Number of participants analyzed = number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 452 | 460
mL | 68 (9) | 8 (9)
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment of the significance level (0.05) was done as a hierarchical approach for hypotheses testing was used; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 60, 95% CI 2-sided [38 to 82], Standard Error of Mean 11

3. Secondary Outcome: COPD Exacerbation Rate (Mild, Moderate or Severe)
Description: Mean rate of COPD exacerbations requiring rescue medication of 3 or more puffs/day on at least 2 consecutive days (=mild COPD exacerbations), or requiring oral or parenteral glucocorticosteroids (=moderate COPD exacerbations), or requiring hospitalization, or leading to death (=severe COPD exacerbations), per patient per year. A COPD exacerbation is an event in the natural course of the disease characterized by a change in the patient's baseline dyspnea, cough and/or sputum beyond day-to-day variability sufficient to warrant a change in management [ATS / ERS 2005].
Time Frame: 24 weeks treatment period
Population: ITT analysis
Measure: Mean (95% Confidence Interval); unit: exacerbations per patient per year
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 466 | 467
exacerbations per patient per year | 1.9 [1.5 to 2.5] | 2.4 [1.9 to 3.1]
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p = 0.1408, Poisson regression — No adjustment of the significance level (0.05) was done as a hierarchical approach for hypotheses testing was used; Rate ratio = 0.79, 95% CI 2-sided [0.58 to 1.08], Standard Error of Mean 0.12

4. Secondary Outcome: Transition Dyspnea Index (TDI) Focal Score
Description: The TDI is a recognized questionnaire to measure dyspnea in an out patient COPD population. At baseline, 3 components of dyspnea, each graded with 4 questions, were asked: - Functional Impairment - Magnitude of Task - Magnitude of Effort At each of the post-randomization visits questions from the TDI were asked related to 3 components: Change in - Functional Impairment - Magnitude of Task - Magnitude of Effort Each question in the TDI is graded from -3 (major deterioration) to +3 (major improvement). This results in a TDI Focal Score ranging from -9 to +9.
Time Frame: Change from baseline over 24 weeks of treatment
Population: ITT analysis. Number of participants analyzed = number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 454 | 460
scores on a scale | 1.2 (0.1) | 1.1 (0.1)
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p = 0.4654, ANCOVA — No adjustment of the significance level (0.05) was done as a hierarchical approach for hypotheses testing was used; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.2 to 0.4], Standard Error of Mean 0.2

5. Secondary Outcome: Shortness of Breath Questionnaire (SOBQ) Total Score
Description: Mean change from baseline during the treatment period in SOBQ. This is a 24-item measure that assesses self-reported shortness of breath while performing a variety of activities of daily living. The questions were administered at visits V0, V2, V3, V4, V5, V6 and Vend to assess the perceived shortness of breath of the patient. For each activity listed in the questionnaire the patient should rate his/her breathlessness on a scale between zero and five, where zero is "not at all breathless" and five is "maximally breathless or too breathless to do the activity".
Time Frame: Change from baseline over 24 weeks of treatment
Population: ITT analysis. Number of participants analyzed = number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 454 | 461
scores on a scale | -0.6 (0.7) | -1.1 (0.7)
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p = 0.5457, ANCOVA — No adjustment of the significance level (0.05) was done as a hierarchical approach for hypotheses testing was used; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.5, 95% CI 2-sided [-1.2 to 2.2], Standard Error of Mean 0.9

ADVERSE EVENTS:
Time Frame: 24 weeks treatment period
Description: The Safety Set was based on all randomized patients who took at least one dose of the investigational drug after randomization.
Arm/Group | Roflumilast | Placebo
Serious Adverse Events (participants affected / at risk) | 36/466 | 42/467
Other Adverse Events (participants affected / at risk) | 165/466 | 143/467
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roflumilast (N=466) | Placebo (N=467)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 11 (11)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Foreign body aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 2 (2) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Arterial restenosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1)
Nodule (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Meningorrhagia (Nervous system disorders) | 1 (1) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Investigation (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Retinitis pigmentosa (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Finger amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roflumilast (N=466) | Placebo (N=467)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 70 (81) | 103 (126) — non-serious
Diarrhoea (Gastrointestinal disorders) | 38 (41) | 15 (16) — non-serious
Nausea (Gastrointestinal disorders) | 25 (26) | 1 (1)
Nasopharyngitis (Infections and infestations) | 33 (39) | 35 (43)
Weight decreased (Investigations) | 39 (39) | 5 (5) — non-serious

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study results may be published and/or presented at scientific meetings. Prior to any submission, all manuscripts/abstracts must be presented to the sponsor for possible comments.